CLINICAL TRIAL: NCT01901484
Title: Intestinal Schistosomiasis in Children Aged 1-5 Years,Morbidity Assessment and the Effect of Praziquantel on Morbidity; Along Lake Victoria Shorelines.
Brief Title: Schistosoma Mansoni Morbidity in Children Aged 1-5 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Allen Nalugwa, Doctor, Makerere University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012162
Record Dates: First submitted 2013-05-30; First posted 2013-07-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Intestinal Schistosomiasis
Keywords: Schistosoma mansoni; morbidity; chemotherapy
MeSH Terms: conditions — Schistosomiasis mansoni; Schistosomiasis | interventions — Praziquantel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug: Praziquantel (Active Comparator): Praziquantel 40mg/Kg - single dose
  Interventions: Drug: Praziquantel
- Praziquantel (Active Comparator): double dose
  Interventions: Drug: Praziquantel

INTERVENTIONS:
Drug: Praziquantel — All the registered S. mansoni infected children aged 1-5 years will be randomly divided into two treatment arms: single and double dose. A second those will be administered after two weeks following the last treatment.

SUMMARY:
This study is about intestinal schistosomiasis, commonly known as bilharzia, in children aged 1-5 years along Lake Victoria shoreline.The children will be screened for S. mansoni and the effects of the disease will be assessed.Children found positive with S. mansoni will be treated with praziquantel and followed up for a year.

DETAILED DESCRIPTION:
The study has three phases: in the first phase (Phase I) a baseline pretreatment schistosomiasis morbidity assessment of children aged 1-5 years will take place. The Kato-Katz technique will be used to detect and enumerate S. mansoni eggs in faecal samples from each participating child. Communities with the highest S. mansoni prevalence and intensity will be chosen and included in the study. In the second phase (Phase II) the S. mansoni positive children will be divided randomly into two intervention groups, single and double dose praziquantel treatment arms. Abdominal ultrasound will be combined with clinical examination to accurately identify hepatosplenomegaly. The sizes of both the liver and spleen will be examined. Anthropometric measurements and Hb for each child will also be recorded. In the last phase (Phase III), the effect of praziquantel on S. mansoni morbidity will be evaluated in all the treated children aged 1-5 years.

ELIGIBILITY:
Inclusion Criteria:

1-5 years

Exclusion Criteria:

<1-5> years

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Presence/absence of organomegaly at Day 0 and 8 months follow-up visits | 2 years

SECONDARY OUTCOMES:
Cure rate at 30 days after treatment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Allen Nalugwa, PhD, Principal Investigator — CHDC-Makerere University; Annette Olsen, PhD, Study Director — University of Copenhagen; Edridah Muheki, PhD, Study Director — Ministry of Health, Vector Control Division; Fred Nuwaha, PhD, Study Director — School of Public Health, Makerere University
Locations (1):
- Child Health & Development Centre, College of Health Sciences , Makerere University, Kampala, Uganda